CLINICAL TRIAL: NCT02832349
Title: Impact of Educational Actions on the Quality Of Life of Epileptic Patients
Acronym: EQOLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15-206
Record Dates: First submitted 2016-07-05; First posted 2016-07-14 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2017-07

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EA group (Educational Actions) (Experimental): Epileptic patients participating to the educational actions program
  Interventions: Other: Educational Actions
- Control group (No Intervention): Epileptic patients with standard follow-up

INTERVENTIONS:
Other: Educational Actions — Individual educational session and 3 group educational sessions (5-6 patients per group) built around the epileptic disease, its treatment and daily life, will constitute the program of EA group.
  Arms: EA group (Educational Actions)

SUMMARY:
The Epilepsy Patient Education (EPE) is very important for the comprehension of the disease and its management. The EPE allows patients and caregivers to acquire together some autonomy and some skills that will help them live better with the disease.The primary objective of this study is to evaluate the impact of a program of educational activities (EA) on the quality of life of epileptic patients measured by the validated scale Quality Of Life in Epilepsy -31 (QOLIE-31).Investigators hope a difference in improving the quality of life score of 25% between the 2 groups.

DETAILED DESCRIPTION:
Introduction:

Epilepsy is a common neurological disease with an estimated annual incidence of 43 cases per 100,000 population in developed countries (McHugh et al;. 2008). It is a chronic disease that can be disabling for the patient and his family. The management of patients with epilepsy must consider the quality of life, improving the quality of life is precisely one of the main objectives of therapeutic education (WHO1996).

Background and rational of the study:

The Epilepsy Patient Education (EPE) is very important for the comprehension of the disease and its management. By offering a better knowledge about the disease, helping the patients to learn how to manage crises and treatments, and especially, how to develop strategies to adapt to specific life situations, the EPE allows patients and caregivers to acquire together some autonomy and some skills that will help them live better with the disease.

Objectives:

The primary objective of this study is to evaluate the impact of a program of educational activities (EA) on the quality of life of epileptic patients measured by the validated scale Quality Of Life in Epilepsy -31 (QOLIE-31).

The secondary objectives are to study the evolution of knowledge of patients, to compare the frequency of crises and seeking care before and after the program, and to study the role of certain characteristics of the patient and his disease on response to the program.

Methodology:

This is a single-center, randomized, open, comparative, and longitudinal study with a duration of approximately 30 months, including 80 patients.

Patients eligible to the study will be screened among epileptic patients followed-up by the neurologists specialized in epilepsy at the University Hospital of Caen. Patients should be major with an epileptic disease diagnosed for at least 6 months without other disabling chronic condition.

Each pre-included patient will receive written information about the study. During the usual visit to the neurologist, a detailed letter of information about the study will be given to the patient and the various criteria will be evaluated. After randomization, patients will be divided into 2 groups: the first (EA group) will be included in the program of educational activities, while the second, control group (C group) will have a "standard" follow-up. An individual educational session and 3 group educational sessions (5-6 patients per group) built around the epileptic disease, its treatment and daily life, will constitute the program of EA group.

Six months after inclusion, during the usual visit, the various criteria will be reassessed with the patient, to evaluate the degree of benefice of EA.

ELIGIBILITY:
Inclusion Criteria:

* Major epileptic patient
* Epilepsy diagnosed for at least 6 months before inclusion

Exclusion Criteria:

* Patient with mental disabilities (patient in an institution or with communication disorders, speech and verbal comprehension)
* Patients with disabling chronic condition other than epilepsy
* Patient consulting for the first time
* Patient whose diagnosis of epilepsy date of less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Score difference at the scale Quality Of Life in Epilepsy -31 (QOLIE-31 ) | Six months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Sophie FONTAINE, Mme, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No